CLINICAL TRIAL: NCT06894381
Title: Characteristics and Results of Patients Treated by Therapeutic Intensification Followed by Autograft of Peripheral Stem Cells and Admitted to Intensive Care and Intensive Care: Single-center Retrospective Analysis
Brief Title: Characteristics and Results of Patients Treated by Therapeutic Intensification
Acronym: AutoREA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9061
Record Dates: First submitted 2024-04-04; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-04

CONDITIONS: Malignant Hemopathy
Keywords: Malignant hemopathy; allogeneic; stem cell; transplantation; chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many studies have focused on patients treated with allogeneic peripheral stem cell transplantation; few studies have until now been carried out to describe the characteristics and results of autografted patients and to attempt to determine possible prognostic factors. However, it is estimated that nearly 5% of autograft patients require MIR care. The investigators therefore wish to conduct a retrospective study including patients treated by therapeutic intensification followed by autograft of hematopoietic stem cells and admitted to the MIR department of the Hautepierre hospital of the University Hospitals of Strasbourg (HUS) within thirty days following initiation of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Gender indifferent
* Admitted to the Intensive Care Unit within thirty days following therapeutic intensification and autograft of peripheral stem cells for the treatment of a hematologic malignancy between 01/01/2013 and 12/31/2022

Exclusion Criteria:

- Subject having expressed his opposition to the reuse of his data for scientific research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) admitted to the Intensive Care Unit within thirty days following therapeutic intensification and autograft of peripheral stem cells for the treatment of a hematologic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the clinical and biological characteristics of patients having therapeutic intensification and autograft of peripheral stem cells for the treatment of hematological malignancy | Thirty days following therapeutic intensification and autograft of peripheral stem cells in treatment of a malignant hematological disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation - CHU de Strasbourg - France, Strasbourg, France